CLINICAL TRIAL: NCT00970281
Title: A Double-Blind Confirmatory Study Comparing Rapid-Acting Intramuscular Olanzapine and Rapid-Acting Intramuscular Placebo in Patients With an Exacerbation of Schizophrenia With Acute Psychotic Agitation
Brief Title: A Study of Olanzapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13333; F1D-JE-RACD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2012-02-22 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 mg Olanzapine (Experimental)
  Interventions: Drug: Rapid-Acting Intramuscular Olanzapine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapid-Acting Intramuscular Olanzapine — Administered by means of intramuscular injection (IM) with the possibility of second 10 milligram (mg) injection 2 to 4 hours after first injection, for a maximum of 2 injections
  Other Names: LY170053; RAIM
  Arms: 10 mg Olanzapine
Drug: Placebo — Administered by means of IM with the possibility of second injection 2 to 4 hours after first injection, for a maximum of 2 injections
  Arms: Placebo

SUMMARY:
The primary objectives of the study is to confirm if the efficacy of intramuscular injection (IM) olanzapine 10 milligrams (mg) in patients with an exacerbation of schizophrenia with acute psychotic agitation is greater than intramuscular placebo by comparing changes from baseline to 2 hours after the first IM injection of agitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision (DSM-IV-TR) criteria for schizophrenia.
* Patients with an exacerbation of schizophrenia with acute psychotic agitation.
* Patients who are hospitalized during the study.
* Patients, or proxy consenters, understand the nature of the study and sign on an informed consent document.
* The investigator or sub-investigator(s) judges that the patients are able to cooperate with all protocol procedures.
* Patients who are considered to be with agitation and appropriate candidates for treatment with intramuscular (IM) medication by the investigator or sub-investigator(s).
* The investigator or sub-investigator(s) believes that it is safe to administer IM olanzapine to the patients in consideration of safety, including the anticholinergic action of IM olanzapine.
* Patients who have a score of 1 or 2 on Agitation-Calmness Evaluation Scale (ACES) before the first IM injection of investigational product.

Exclusion Criteria:

* Patients whose Global Assessment of Functioning (GAF) score is less than or equal to 40 within last 1 year before informed consent.
* Patients with defect.
* Patients whose agitation continues more than 2 weeks before informed consent.
* Patients who were previously treated with antipsychotics and were considered by the investigator or sub-investigator(s) to be treatment-resistant to antipsychotics.
* Patients who were treated by oral olanzapine at a dose of more than 20 milligrams (mg) for more than 4 weeks but did not improve.
* Patient who have a history of participation in clozapine trials or treatment with clozapine.
* Patients who have co-morbidity of mental retardation and personality disorder.
* Patients whose agitation is possibly due to brain lesions such as (but not limited to) head injury, stroke, brain breeding, and cerebral infection.
* Patients with sub-stupor or stupor.
* One or more seizures without a clear and resolved etiology. However, if the patient has had one or more seizures in the past with an identifiable etiology, and that etiology has been resolved, the patient may be entered.
* Patients who have a history of DSM-IV-TR substance (except caffeine and nicotine) abuse within the past 30 days or substance dependence within the past 6 months before informed consent. Or patients who have a history of using illegal drug.
* Patients whose agitation is caused by substance abuse or neurologic conditions, in the opinion of the investigator or sub-investigator(s).
* Patients who have a diagnosis of Parkinson's disease or dementia.
* Patients who are actively suicidal (at high risk for suicide attempt) in the opinion of the investigator or sub-investigator(s).
* Patients with inadequately controlled diabetes, or patients whose treatment for diabetes has been changed within 4 weeks before the first IM injection of the investigational product. The investigator's discretion will supersede even if the patients do not meet the above criteria for concurrent diabetes.
* Patients who have received haloperidol decanoate fluphenazine decanoate, or fluphenazine enanthate within 8 weeks before the first IM injection of investigational product.
* Patients who have received risperidone long-acting injection within 12 weeks before the first IM injection of investigational product.
* Patients who have a history of receiving injectable depot antipsychotics other than haloperidol decanoate, fluphenazine decanoate, fluphenazine enanthate and risperidone long-acting injection.
* Patients who have received antipsychotics or other prohibited concomitant medicines within 2 hours before the first IM injection of investigational product.
* Patients who have received benzodiazepines within 4 hours before the first IM injection of investigational product.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time(UTC/GMT-5hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

REFERENCES:
- [Derived] Katagiri H, Fujikoshi S, Suzuki T, Fujita K, Sugiyama N, Takahashi M, Gomez JC. A randomized, double-blind, placebo-controlled study of rapid-acting intramuscular olanzapine in Japanese patients for schizophrenia with acute agitation. BMC Psychiatry. 2013 Jan 11;13:20. doi: 10.1186/1471-244X-13-20. PMID 23311957

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg Olanzapine: Administered by means of intramuscular injection (IM) with the possibility of second 10 milligram (mg) injection 2 to 4 hours after first injection, for a maximum of 2 injections.
- Placebo: Administered by means of IM injection with the possibility of second injection 2 to 4 hours after first injection, for a maximum of 2 injections.
Period: Overall Study
Arm/Group | 10 mg Olanzapine | Placebo
Started | 46 | 45
Full Analysis Set | 45 (1 participant in the olanzapine arm discontinued before the first intramuscular (IM) injection.) | 45
Completed | 44 | 29
Not Completed | 2 | 16
Not completed — Lack of Efficacy | 1 | 14
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Olanzapine | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.7) | 47.0 (12.1) | 46.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  Japan | 45 | 45 | 90
Diabetes Mellitus Status [Number; unit: participants]
  Diabetes Mellitus - Yes | 3 | 3 | 6
  Diabetes Mellitus - No | 42 | 42 | 84
Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision Diagnosis Status [Number; unit: participants] — Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision (DSM-IV-TR) diagnosis status.
  participants
    Catatonic | 0 | 2 | 2
    Disorganized | 4 | 3 | 7
    Paranoid | 40 | 40 | 80
    Undifferentiated | 1 | 0 | 1
    Residual | 0 | 0 | 0
Pre-therapy Antipsychotic Usage [Number; unit: participants]
  Yes (>=1000 milligrams [mg]) | 12 | 11 | 23
  Yes (<1000 mg) | 27 | 30 | 57
  No | 6 | 4 | 10
Age at Onset [Mean (Standard Deviation); unit: years] | 24.7 (9.4) | 27.2 (9.3) | 25.9 (9.4)
Agitation-Calmness Evaluation Scale (ACES) Score [Mean (Standard Deviation); unit: units on a scale] — The ACES differentiates agitation, calmness, and sleep-state, using a 9-point scale: 1 (Marked Agitation) to 9 (Unarousable).
  units on a scale | 1.6 (0.5) | 1.6 (0.5) | 1.6 (0.5)
Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) Total Score [Mean (Standard Deviation); unit: units on a scale] — Measures excitability and consists of the following 5 items from the PANSS: Excitement, Hostility, Tension, Uncooperativeness, and Poor Impulse Control. Each item is rated on a scale from 1 (absent) to 7 (extreme). The sum of the 5 items is defined as the PANSS-EC total score which ranges from 5 to 35.
  units on a scale | 23.5 (6.1) | 23.2 (4.9) | 23.4 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) Total Score up to 2 Hours After the First Intramuscular (IM) Injection
Description: Measures excitability and consists of the following 5 items from the PANSS: Excitement, Hostility, Tension, Uncooperativeness, and Poor Impulse Control. Each item is rated on a scale from 1 (absent) to 7 (extreme). The sum of the 5 items is defined as the PANSS-EC total score which ranges from 5 to 35.
Time Frame: Baseline, up to 2 hours after first IM injection
Population: Participants with a baseline and a value at the time, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
units on a scale | -9.2 (4.5) | -2.8 (5.6)
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Sample size of at least 45 participants per group was necessary to verify decreases in PANSS-EC total score were significantly greater in olanzapine group than placebo group using a t-test with a power of 90% and a 2-sided significance level of 5%; Test type: Superiority or Other; p < 0.001, ANOVA — The p-value was based on an analysis of variance (ANOVA) model that included treatment and site as a factor

2. Secondary Outcome: Change From Baseline in PANSS-EC Total Score up to 90 Minutes After the First Intramuscular (IM) Injection
Description: as for outcome 1
Time Frame: Baseline, 15 minutes, 30 minutes, 60 minutes, and 90 minutes after the first injection
Population: Full analysis set (FAS): All randomized participants administered at least 1 intramuscular (IM) injection of the investigational product with at least 1 observation after the first IM injection, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
units on a scale
  0.25 hour after First IM Injection | -2.4 (2.9) | -1.0 (3.1)
  0.50 hour after First IM Injection | -5.0 (3.6) | -1.9 (4.6)
  1 hour after First IM Injection | -7.3 (4.9) | -3.0 (5.2)
  1.5 hour after First IM Injection | -8.2 (4.7) | -2.7 (5.0)
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.009, ANOVA — This is the p-value for 0.25 hour after first IM injection
Statistical Analysis 2: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — This is the p-value for the 0.50 hour after first IM injection
Statistical Analysis 3: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — This is the p-value for the 1 hour after first IM injection
Statistical Analysis 4: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — This is the p-value for the 1.5 hour after first IM injection

3. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC) Total Score up to 24 Hours After the First Intramuscular (IM) Injection
Description: as for outcome 1
Time Frame: Baseline, up to 24 hours after first IM injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
units on a scale | -5.6 (5.8) | -2.8 (6.4)
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, ANOVA

4. Secondary Outcome: Percentage of Participants With 40% or Greater Percent Decrease in the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC) Total Score up to 2 Hours After the First Intramuscular (IM) Injection
Description: as for outcome 1
Time Frame: Up to 2 hours after the first (IM) injection
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
percentage of participants | 40.0 | 13.6
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Scores of 4 to 7 in the Agitation-Calmness Evaluation Scale (ACES) Score up to 24 Hours After the First Intramuscular (IM) Injection
Description: The ACES differentiates agitation, calmness, and sleep-state, using a 9-point scale: 1 (Marked Agitation) to 9 (Unarousable). Scores of 4 (Normal) to 7 (Marked Calmness) were used for this outcome measure.
Time Frame: up to 24 hours after the first IM injection
Population: Participants having a post-baseline measure, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
percentage of participants
  0.5 hour after First IM Injection | 24.4 | 11.4
  1 hour after First IM Injection | 31.1 | 15.9
  1.5 hours after First IM Injection | 40.0 | 13.6
  2 hours after First IM Injection | 40.0 | 13.6
  24 hours after First IM Injection | 28.9 | 15.9
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.167, Fisher Exact — This is the p-value for the 0.5 hour after the first IM injection
Statistical Analysis 2: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.134, Fisher Exact — This is the p-value for the 1 hour after the first IM injection
Statistical Analysis 3: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact — This is the p-value for the 1.5 hour after the first IM injection
Statistical Analysis 4: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact — This is the p-value for the 2 hours after the first IM injection
Statistical Analysis 5: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.204, Fisher Exact — This is the p-value for the 24 hours after the first IM injection

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Extrapyramidal Symptoms Based on the Drug Induced Extrapyramidal Symptoms Scale (DIEPSS) Score up to 24 Hours After the First Intramuscular (IM) Injection
Description: Assesses extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms; 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). Total points of 8 items are defined as DIEPSS total (0 to 32 points). Items for assessment of individual symptoms are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Parkinsonism is assessed by total points of items 1 to 5; akathisia, dystonia and dyskinesia are assessed by points given to corresponding items (item 6, item 7, and item 8, respectively).
Time Frame: Up to 24 hours after the first IM injection
Population: Participants with an abnormal value at post-baseline, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Olanzapine | Placebo
Number analyzed (Participants) | 45 | 44
percentage of participants
  Parkinsonism (N=43, 44) | 4.7 | 6.8
  Akathisia (N=43, 45) | 0.0 | 0.0
  Dystonia (N=44, 45) | 0.0 | 0.0
  Dyskinesia (N=44, 45) | 0.0 | 0.0
Statistical Analysis 1: Comparison: 10 mg Olanzapine vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — This is the p-value for Parkinsonism

ADVERSE EVENTS:
Arm/Group | 10 mg Olanzapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 13/45 | 6/45
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg Olanzapine (N=45) | Placebo (N=45)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days